CLINICAL TRIAL: NCT06935149
Title: Detecting Liver Metastatic Lesions in Patients of Colorectal Cancer With Novel Precise Imaging Tools
Brief Title: Detecting Colorectal Cancer With Liver Metastatic Lesions Using Novel Precise Imaging Tools
Acronym: PSMA
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Primo Biotechnology Co., Ltd (Industry)
Collaborators: Kaohsiung Chang Gung Memorial Hospital,Taiwan (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: PB012Co
Record Dates: First submitted 2025-04-11; First posted 2025-04-20 (Actual); Last update posted 2025-04-24 (Actual); Status verified 2025-04

CONDITIONS: Liver Metastasis Colon Cancer
Keywords: Liver metastasis; PSMA; PET
MeSH Terms: interventions — PSMA-BCH

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PSMA-PET (Experimental)
  Interventions: Drug: 18-PSMA

INTERVENTIONS:
Drug: 18-PSMA — Intravenous push 4 MBq/kg per patient (for a 70 kg patient, 280 MBq of [18F]FPSMA needs to be intravenously injected), and the maximum dose cannot exceed 400 MBq. After the injection of [18F]FPSMA, intravenous flushing was performed with 20 ml of normal saline.

SUMMARY:
This study will demonstrate the diagnostic utility of PSMA PET among patients with CRC with liver metastasis.

ELIGIBILITY:
Main inclusion criteria:

1. The participants can voluntarily sign informed consent forms
2. The participants are male/female over 20 years old.
3. The participant is currently undergoing cancer staging based on the previous pathological diagnosis of colorectal cancer
4. The participants are confirmed liver metastasis by CT, abdominal ultrasound, MRI, and FDG PET/CT within 30 days before receiving PSMA-PET/CT.
5. WHO performance status ≦ 2 points
6. The participants can lie on table for two hours during PSMA-PET/CT scanning.

Main exclusion criteria: To improve the accurate interpretation of PMSA-PET imaging and reduce the occurrence of related-drug adverse events, the participants will be excluded by following below criteria.

1. The colorectal cancer participants was diagnosed other organs metastases with multiple organ metastases not only the liver.
2. The colorectal cancer participants have undergone any treate after diagnosis of liver metastasis.
3. The participants have suffered from liver dysfunction such as AST/ALT ratio >2、total bilirubin >1.5 mg/dL within 6 months.
4. The participants suffered stage IV chronic kidney disease (eGFR<30 mL/min/1.73 m2) within 6 months.
5. The participants suffered acute kidney injury within 6 months.
6. The participants suffered trauma or fracture.
7. The participants are allergic to any radiopharmaceutical or imaging agent.
8. The participants are history of claustrophobia or are inability to remain quiet during the examination.

Ages: 20 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Estimated)
Dates: Start 2025-05-01 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
PSMA positive detection rate is defined as the rate that is detected positive lesion at the same location/region between [18F]FPSMA-1007 PET/CT (60- minute images) and reference standard. | 14 days

IPD SHARING:
Plan to Share IPD: No